CLINICAL TRIAL: NCT07091773
Title: A Clinical Trial to Evaluate the Safety and Effectiveness of "OLIZ," a Combined Wavelength Photobiomodulation Medical Device, for Surgical Site Pain Relief in Patients Who Have Undergone Total Knee Arthroplasty (TKA) : A Multicenter, Controlled, and Randomized Clinical Trial
Brief Title: A Clinical Trial to Evaluate the Safety and Effectiveness of OLIZ, a Photobiomodulation Medical Device for Surgical Site Pain Relief in Patients After Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LTBIO Co., Ltd. (Industry)
Collaborators: Inje University (Other); InjeUniversityIlsanPaikHospital (Unknown); Gangnam Severance Hospital (Other); National Medical Center, Seoul (Other); National Health Insurance Service Ilsan Hospital (Other); Korea University Anam Hospital (Other); Samsung Medical Center (Other); The Catholic University of Korea Uijeongbu St.Marys Hostpial (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT_Knee_Pain-02
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain Management During Rehabilitation in Patients Undergoing Total Knee Arthroplasty
Keywords: photobiomodualtion; Total knee arthroplasty; Postoperative pain; Rehabilitation; Pain management
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Statistical analyst responsible for data analysis is masked from randomization assignments and clinical data access until database lock completion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OLIZ Photobiomodulation Treatment (Experimental): Participants will receive photobiomodulation therapy using the OLIZ device, which delivers dual-wavelength light therapy (red and near-infrared spectrum) to the surgical site. Treatment will begin within 3 days post-surgery and continue according to the postoperative care protocol. The OLIZ device targets cellular pathways involved in inflammation reduction, microcirculation enhancement, and tissue repair to manage postoperative pain and promote recovery in total knee arthroplasty patients.
  Interventions: Device: OLIZ Photobiomodulation Device
- Standard care control (No Intervention): Participants will receive standard postoperative care including conventional pain management protocols without photobiomodulation therapy. All other aspects of postoperative care will be identical to the treatment group.

INTERVENTIONS:
Device: OLIZ Photobiomodulation Device — OLIZ device utilizes dual-wavelength technology combining specific red (660nm) and near-infrared (850nm) light parameters optimized for post-surgical tissue healing. The device features controlled power density, precise treatment duration protocols, and targeted application to knee arthroplasty surgical sites. Treatment parameters include specific irradiance levels, treatment session duration of 15 minutes, and 3 times of daily application frequency designed.
  Arms: OLIZ Photobiomodulation Treatment

SUMMARY:
A Clinical Trial to Evaluate the Safety and Effectiveness of OLIZ, a Photobiomodulation Medical Device for Surgical Site Pain Relief in Patients After Total Knee Arthroplasty

DETAILED DESCRIPTION:
This multicenter, controlled, randomized clinical trial is designed to evaluate the safety and effectiveness of "OLIZ," a medical device that utilizes combined-wavelength photobiomodulation (PBM) therapy, for relieving postoperative pain at the surgical site in patients undergoing total knee arthroplasty (TKA).

Photobiomodulation therapy employs specific wavelengths of light to modulate biological processes at the cellular level, such as reducing inflammation, enhancing microcirculation, and promoting tissue repair. OLIZ delivers dual-wavelength light in the red and near-infrared spectrum, targeting key cellular pathways involved in postoperative pain and recovery.

Participants in the study will be randomly assigned to receive either the active PBM treatment using OILZ or a control intervention. Treatment will begin within 3 days after surgery and continue for a defined period based on the postoperative care protocol. VAS, WOMAC, and recovery metrics will be monitored at multiple time points during the inpatient stay and follow-up period.

The study also aims to assess the safety of repeated PBM exposure in a post-surgical setting by evaluating local and systemic adverse events. Through this trial, investigators seek to generate robust clinical evidence to support the use of OLIZ as a non-pharmacologic modality for pain management and recovery enhancement in TKA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥19 years and <80 years at the time of consent
2. Radiographic evidence (X-ray) within 24 weeks prior to total knee arthroplasty (TKA) showing Kellgren-Lawrence (KL) grade 4 in the surgical knee
3. Surgical site pain confirmed as a visual analog scale (VAS) score ≥50.0
4. Willingness to refrain from any treatments not permitted by the study protocol, aside from concomitant medications or therapies allowed during the study period
5. Voluntary participation in the clinical trial with written informed consent provided after being fully informed of the study procedures
6. Willingness and ability to comply with the requirements of the clinical trial protocol

Exclusion Criteria:

Subjects will be excluded from this clinical trial if they meet any of the following criteria:

1. History of surgery, other than total knee arthroplasty, in the area of the knee joint being evaluated (or scheduled for surgery).*

   *Includes total/partial knee arthroplasty, knee cartilage surgery, knee ligament reconstruction, autologous chondrocyte implantation, knee fracture surgery, knee synovectomy/loose body removal, patellar reconstruction, patellar realignment, bursectomy, synovectomy, etc.
2. History of using steroids or immunosuppressants at the time of screening, meeting one or more of the following:

   Immunosuppressants (e.g., cyclosporin A or azathioprine) within 6 weeks.

   Oral steroids or antidepressants within 4 weeks.

   Intra-articular injection* into the target knee joint within 12 weeks.

   *Includes steroids, hyaluronic acid, polynucleotide, PDRN (polydeoxyribonucleotide), etc.
3. Determined to be unable to wear the device due to one or more of the following:

   Individuals with photosensitive skin.

   Individuals taking medications that may cause light sensitivity (refer to the precautions of the medication being taken).

   Individuals with sensitive skin due to an allergic constitution.

   Individuals with implanted electronic medical devices.
4. Meeting one or more of the following physical examination or laboratory test results at the time of screening:

   Fever exceeding 37.8°C.

   PT (INR) or aPTT ≥ 1.5 x ULN (upper limit of normal).

   Serum creatinine > 1.5 x ULN.

   AST or ALT ≥ 2.0 x ULN.

   (Only for those with a history of diabetes) Glycosylated hemoglobin (HbA1c) > 11%.
5. History of one or more of the following medical conditions or diseases confirmed at the time of screening:

   Secondary osteoarthritis such as rheumatoid arthritis, Paget's disease, or gouty arthritis (however, traumatic osteoarthritis is permitted for enrollment).

   History of cardiac disease such as myocardial infarction or congestive heart failure.

   Uncontrolled hypertension (SBP > 160 mmHg or DBP > 100 mmHg).

   History of uncontrolled endocrine abnormalities or diseases (e.g., thyroid disease, parathyroid disease, pituitary disease).

   Immune system-related diseases (e.g., infectious diseases, systemic lupus erythematosus).

   History of malignancy within the last 5 years (however, individuals with a history of basal cell or squamous cell skin cancer and non-invasive carcinomas are eligible to participate in the clinical trial only if adequately treated).
6. Pregnant or lactating women.
7. Women of childbearing potential who do not agree to use medically acceptable birth control methods* during the clinical trial period.

   *Hormonal contraception, intrauterine devices, tubal ligation, double barrier methods (combined use of barrier methods such as male condoms, female condoms, cervical caps, diaphragms, contraceptive sponges), or a single barrier method combined with spermicide.
8. Currently participating in another clinical trial or having participated in another clinical trial within 30 days prior to the screening date.
9. Any other case where, in the investigator's judgment, participation in the clinical trial is deemed inappropriate due to ethical reasons or potential impact on the clinical trial results.

   -

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in VAS Pain Score | Baseline and 11 weeks post-baseline
  Primary efficacy endpoint measuring the change in pain intensity using Visual Analog Scale from baseline to 11 weeks post-baseline. VAS scores range from 0mm (no pain) to 100mm (worst possible pain).

SECONDARY OUTCOMES:
Change in VAS Pain Score at 5 weeks | Baseline and 5 weeks post-baseline
  Secondary efficacy endpoint measuring the change in pain intensity using Visual Analog Scale from baseline to 5 weeks post-baseline. VAS scores range from 0mm (no pain) to 100mm (worst possible pain).
Change from baseline in WOMAC total score at Week 5 and Week 11 | Baseline, Week 5, and Week 11 post-surgery
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) total score assesses pain, stiffness, and physical function. The change from baseline to Week 5 and Week 11 post-surgery will be measured to evaluate the effectiveness of the intervention on postoperative recovery.
Change from baseline in knee joint range of motion (ROM) at Week 5 and Week 11 | Baseline, Week 5, and Week 11 post-surgery
  Range of motion (ROM) of the knee joint, including flexion and extension, will be measured using a goniometer. The change in ROM from baseline to Week 5 and Week 11 post-surgery will be assessed to evaluate the effect of the intervention on functional recovery.
Change from baseline in the cumulative dose of rescue and prescribed analgesic medications at Week 5 and Week 11 | Baseline, Week 5, and Week 11 post-surgery
  The total cumulative dose (in mg) of prescribed and rescue analgesic medications (e.g., acetaminophen, NSAIDs, opioids) taken by each participant will be recorded. The change from baseline to Week 5 and Week 11 will be assessed to evaluate the effect of the intervention on the need for pharmacologic pain management.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Wook Nha, M.D., Ph.D, Principal Investigator — Inje University Ilsan Paik Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality concerns that cannot be adequately addressed with de-identification methods, particularly given the small sample size and unique characteristics of the study population.